CLINICAL TRIAL: NCT04892472
Title: EF-36/Keynote B36: A Pilot, Randomized, Open-label Study of Tumor Treating Fields (TTFields, 150 kHz) Concomitant With Pembrolizumab for First Line Treatment of Advanced or Metastatic Non-small Cell Lung Cancer
Acronym: KEYNOTE B36
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Phase 2 study terminated due to insufficient enrollment and was not based on safety concerns. Novocure is enrolling a new Phase 3 study of TTFields as a first line treatment for advanced/metastatic NSCLC (NCT06216301).
Sponsor: NovoCure GmbH (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: NovoCure Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EF- 36; KEYNOTE-B36 (Other: Merck Sharp & Dohme Corp)
Record Dates: First submitted 2021-05-13; First posted 2021-05-19 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; NSCLC; Advanced non-small cell lung cancer; Metastatic non-small cell lung cancer; Immunotherapy; PDL-1 positive; Treatment; Minimal toxicity; TTFields; Tumor Treating Fields; Novocure; Pembrolizumab; Merck
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Arm 1: Treatment Group (Experimental): Pembrolizumab (MK-3475) and TTFields
  Interventions: Device: NovoTTF-200T; Drug: Pembrolizumab (MK-3475) 200 mg
- Arm 2: Control Group (Experimental): Pembrolizumab (MK-3475)
  Interventions: Drug: Pembrolizumab (MK-3475) 200 mg

INTERVENTIONS:
Device: NovoTTF-200T — All patients enrolled in this group will receive TTFields treatment, delivered for at an average of least 18 hours a day using NovoTTF-200T concomitant with pembrolizumab, a standard immunotherapy agent, which is delivered intravenously.
  Arms: Arm 1: Treatment Group
Drug: Pembrolizumab (MK-3475) 200 mg — Pembrolizumab (MK-3475) 200 mg every 3 weeks (Q3W)

SUMMARY:
This is a multicenter, randomized, open-label study of Tumor Treating Fields (TTFields) at 150 kHz to the thorax using the NovoTTF-200T System with IV pembrolizumab in subjects previously untreated for advanced or metastatic, PD-L1 positive non-small cell lung cancer (NSCLC). The primary objective is to evaluate the progression-free survival (PFS) by RECIST 1.1 in subjects with TPS ≥1 percent, 1L metastatic/current advanced NSCLC treated with TTFields concomitant with pembrolizumab compared to those treated with pembrolizumab alone.

The device is an experimental, portable, battery operated device for chronic administration of alternating electric fields (termed TTFields) to the region of the malignant tumor, by means of surface, insulated electrode arrays.

DETAILED DESCRIPTION:
TTFields have demonstrated significant activity in vitro and in NSCLC pre-clinical models, both as a single modality treatment and concomitant with chemotherapies and PD-1 inhibitors. TTFields have demonstrated synergistic activity when administered alongside taxanes; while TTFields used concomitantly with PD-1 inhibition have shown additive effects.

In a pilot study, 42 advanced stage NSCLC patients, who had tumor progression after at least one line of prior chemotherapy, received pemetrexed together with TTFields (150 kHz) applied to the chest and upper abdomen until disease progression. The combination was well tolerated and the only device-related adverse event was mild to moderate contact dermatitis. Efficacy endpoints were remarkably high compared to historical data for pemetrexed alone.

Preclinical models have been used to assess the potency of TTFields concomitant with checkpoint inhibition. In an in vivo experiment, C57Bl/6 mice had LLC-1 cells injected directly into the lungs. TTFields were applied to the mouse lungs for 7 days in parallel to I.P. injections of anti-PD-1. Concomitant TTFields and anti-PD-1 treatments led to a significant decrease in tumor volume compared to control mice and to mice treated with anti-PD-1 alone. The concomitant treatments also resulted in an increase in the percentage of tumor-infiltrating leukocytes (CD45+). Specifically, there was a significantly higher frequency of macrophages (CD45+/CD11b+/F4/80+) and dendritic cells (CD45+/CD11c+) in tumors from mice that were concomitantly treated with TTFields and anti-PD-1. Concomitant therapy upregulated PD-1 expression on macrophages and dendritic cells in mice, suggesting an adaptive immune response to control the inflammation caused by the treatment. Additionally, cytotoxic T-cells isolated from tumors treated with TTFields and anti-PD-1 demonstrated increased production of IFN-γ. Overall, these findings imply that concomitant TTFields and anti-PD-1 therapy enhanced the immune response, which led to better management of the tumor.

The study will enroll 100 patients, whose tumors are classified as TPS>1% and in whom EGFR or ALK-directed therapy is not indicated, for examination of the effectiveness and safety of TTFields concomitant with pembrolizumab.

In addition, all patients must meet all eligibility criteria.

After a Screening Phase of up to 28 days, subjects will be enrolled to receive TTFields (150 kHz) to the thorax using the NovoTTF-200T device for an average of 18 hours a day concomitant with pembrolizumab 200 mg IV every 3 weeks, or pembrolizumab alone. Each subject will participate in the study for approximately 2 years from the time the subject signs the Informed Consent Form (ICF) through the final contact.

Treatment with TTFields and pembrolizumab will continue for 24 months (TTFields) and until either: (1) 35 study treatments have been administered (pembrolizumab), (2) there is documented disease progression (per iRECIST criteria), (3) unacceptable adverse event(s), (4) intercurrent illness that prevents further administration of treatment, (5) investigator's decision to withdraw the subject, (6) subject withdraws consent, (7) pregnancy of the subject, (8) non-compliance with study treatment or procedure requirements, or (9) administrative/Sponsor decisions.

In case of discontinuation of either of the study treatments due to reasons other than disease progression, the remaining treatment should continue until disease progression or 24 months (TTFields) / 35 cycles (pembrolizumab).

If an alternative anticancer therapy is initiated, the patient will be removed from the study.

Subjects who discontinue all study treatments prior to disease progression will be monitored for disease status in the Observation Phase until: (1) disease progression is confirmed by the site, (2) a non-study cancer treatment is initiated, (3) consent is withdrawn, or (4) the subject is lost to follow-up. Subjects will have post-treatment monthly follow-up by telephone for disease status until death, withdrawing consent, becoming lost to follow-up, or end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of stage III or metastatic NSCLC without EGFR sensitizing mutation or ALK translocation
* Age ≥ 22 years
* Have a PD-L1 positive (TPS≥1%) tumor by local laboratory assessment
* Have evaluable (measureable or non-measureable) disease in thorax per RECIST 1.1
* ECOG performance status of 0 to 1
* Have not received prior treatments for metastatic or current advanced NSCLC. Palliative treatment is allowed and subjects who received adjuvant, neoadjuvant chemotherapy or chemoradiotherapy with curative intent for non-metastatic disease are eligible if therapy completed at least 12 months prior to the development of metastatic or current advanced disease.
* Life expectancy of at least 3 months
* Able to operate the NovoTTF-200T device

Exclusion Criteria:

* Has known active or untreated CNS metastases and/or carcinomatous meningitis
* Has an EGFR sensitizing mutation and/ or ALK translocation
* Can be treated with curative intent with either surgical resection and/or chemoradiation
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or an agent directed to another stimulatory or co-inhibitory T cell receptor within the past 12 months
* Has received prior systemic anti-cancer therapy for metastatic or current advanced NSCLC (palliative radiotherapy is allowed)
* Being unable to operate the NovoTTF-200T device independently or with the help of a caregiver
* Pregnancy or breastfeeding
* Received live vaccine in the past 30 days or had major surgery in the last 3 weeks
* Is expected to require any other form of systemic or localized antineoplastic therapy while on study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 24 months
  PFS will be measured from the date of enrollment to date of progression (in months) based on RECIST 1.1 criteria. The analysis will include stratification by PD-L1 expression, TPS≥1-49% and TPS≥50%, as a secondary outcome.

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
  Survival will be measured from date of enrollment until date of death. The analysis will include patients with PD-L1 expression TPS≥1-49 percent and TPS≥50 percent
Objective Response Rate (ORR) | 24 months
  Percentage of patients who have a partial or complete response to therapy based on RECIST 1.1 criteria
Duration of response (DOR) | 24 months
  The analysis will be defined as the time from response to progression/death (P/D) based on RECIST 1.1 criteria
Disease control rate (DCR) | 18 weeks
  Will be defined as the percentage of patients with advanced or metastatic cancer who have achieved complete response (CR), partial response (PR), and stable disease (SD) by RECIST 1.1 at 18 weeks
Safety and Tolerability: adverse events (AEs) | 24 months
  Will be defined as the incidence, frequency and severity of adverse events (AEs) noted in patients treated.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Central Alabama Research, Birmingham, Alabama
  - Palo Verde Cancer Specialists, Glendale, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - Long Beach Memorial Medical Center, Long Beach, California
  - UCHealth Memorial Hospital, Colorado Springs, Colorado
  - Cancer Care of North Florida, Lake City, Florida
  - Miami Cancer Insititute - Baptist Health South Florida, Miami, Florida
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Franciscan St. Francis Health Indianapolis, Indianapolis, Indiana
  - Saint Elizabeth Healthcare, Edgewood, Kentucky
  - Baptist Health Oncology Research, Lexington, Kentucky
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Cancer and Leukemia Center, Sterling Heights, Michigan
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - OptumCare Cancer Care, Las Vegas, Nevada
  - Arnot Ogen Medical Center - Falck Cancer Center, Elmira, New York
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Gabrail Cancer Research Center, Canton, Ohio
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Texas Oncology - Sammons Cancer Center, Dallas, Texas
  - : The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee SX, Wong ET, Swanson KD. Mitosis Interference of Cancer Cells by NovoTTF-100A Causes Decreased Cellular Viability. Cancer Res. 2013;73; 709. http://cancerres.aacrjournals.org/content/73/8%7B_%7DSupplement/709.abstract.
- [Background] Bomzon Z, Urman N, Wenger C, et al. Transducer array layout optimization for treating lung-based tumors with TTFields. J Clin Oncol. 2015;33(suppl; abstr e18503). http://meetinglibrary.asco.org/content/147908-156.
- [Background] Pless M, Droege C, von Moos R, Salzberg M, Betticher D. A phase I/II trial of Tumor Treating Fields (TTFields) therapy in combination with pemetrexed for advanced non-small cell lung cancer. Lung Cancer. 2013;81(3):445-450. doi:10.1016/j.lungcan.2013.06.025 17. Hanna N, Shepherd FA, Fossella F V, et al. Randomized phase III trial of pemetrexed versus docetaxel in patients with non-small-cell lung cancer previously treated with chemotherapy. J Clin Oncol. 2004;22(9):1589-1597. doi:10.1200/JCO.2004.08.163
- [Result] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Result] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Result] Giladi M, Schneiderman RS, Voloshin T, Porat Y, Munster M, Blat R, Sherbo S, Bomzon Z, Urman N, Itzhaki A, Cahal S, Shteingauz A, Chaudhry A, Kirson ED, Weinberg U, Palti Y. Mitotic Spindle Disruption by Alternating Electric Fields Leads to Improper Chromosome Segregation and Mitotic Catastrophe in Cancer Cells. Sci Rep. 2015 Dec 11;5:18046. doi: 10.1038/srep18046. PMID 26658786
- [Result] Pless M, Weinberg U. Tumor treating fields: concept, evidence and future. Expert Opin Investig Drugs. 2011 Aug;20(8):1099-106. doi: 10.1517/13543784.2011.583236. Epub 2011 May 9. PMID 21548832
- [Result] Mun EJ, Babiker HM, Weinberg U, Kirson ED, Von Hoff DD. Tumor-Treating Fields: A Fourth Modality in Cancer Treatment. Clin Cancer Res. 2018 Jan 15;24(2):266-275. doi: 10.1158/1078-0432.CCR-17-1117. Epub 2017 Aug 1. PMID 28765323
- [Result] Giladi M, Weinberg U, Schneiderman RS, Porat Y, Munster M, Voloshin T, Blatt R, Cahal S, Itzhaki A, Onn A, Kirson ED, Palti Y. Alternating electric fields (tumor-treating fields therapy) can improve chemotherapy treatment efficacy in non-small cell lung cancer both in vitro and in vivo. Semin Oncol. 2014 Oct;41 Suppl 6:S35-41. doi: 10.1053/j.seminoncol.2014.09.006. Epub 2014 Sep 8. PMID 25213867
- [Result] Voloshin T, Kaynan N, Davidi S, Porat Y, Shteingauz A, Schneiderman RS, Zeevi E, Munster M, Blat R, Tempel Brami C, Cahal S, Itzhaki A, Giladi M, Kirson ED, Weinberg U, Kinzel A, Palti Y. Tumor-treating fields (TTFields) induce immunogenic cell death resulting in enhanced antitumor efficacy when combined with anti-PD-1 therapy. Cancer Immunol Immunother. 2020 Jul;69(7):1191-1204. doi: 10.1007/s00262-020-02534-7. Epub 2020 Mar 6. PMID 32144446
- [Result] Kirson ED, Giladi M, Gurvich Z, Itzhaki A, Mordechovich D, Schneiderman RS, Wasserman Y, Ryffel B, Goldsher D, Palti Y. Alternating electric fields (TTFields) inhibit metastatic spread of solid tumors to the lungs. Clin Exp Metastasis. 2009;26(7):633-40. doi: 10.1007/s10585-009-9262-y. Epub 2009 Apr 23. PMID 19387848
- [Result] Bomzon Z, Urman N, Wenger C, Giladi M, Weinberg U, Wasserman Y, Kirson ED, Miranda PC, Palti Y. Modelling Tumor Treating Fields for the treatment of lung-based tumors. Annu Int Conf IEEE Eng Med Biol Soc. 2015;2015:6888-91. doi: 10.1109/EMBC.2015.7319976. PMID 26737876
- [Result] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Result] Kirson ED, Schneiderman RS, Dbaly V, Tovarys F, Vymazal J, Itzhaki A, Mordechovich D, Gurvich Z, Shmueli E, Goldsher D, Wasserman Y, Palti Y. Chemotherapeutic treatment efficacy and sensitivity are increased by adjuvant alternating electric fields (TTFields). BMC Med Phys. 2009 Jan 8;9:1. doi: 10.1186/1756-6649-9-1. PMID 19133110
- [Result] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225
- [Result] Taphoorn MJB, Dirven L, Kanner AA, Lavy-Shahaf G, Weinberg U, Taillibert S, Toms SA, Honnorat J, Chen TC, Sroubek J, David C, Idbaih A, Easaw JC, Kim CY, Bruna J, Hottinger AF, Kew Y, Roth P, Desai R, Villano JL, Kirson ED, Ram Z, Stupp R. Influence of Treatment With Tumor-Treating Fields on Health-Related Quality of Life of Patients With Newly Diagnosed Glioblastoma: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2018 Apr 1;4(4):495-504. doi: 10.1001/jamaoncol.2017.5082. PMID 29392280
- [Result] Vogelzang NJ, Rusthoven JJ, Symanowski J, Denham C, Kaukel E, Ruffie P, Gatzemeier U, Boyer M, Emri S, Manegold C, Niyikiza C, Paoletti P. Phase III study of pemetrexed in combination with cisplatin versus cisplatin alone in patients with malignant pleural mesothelioma. J Clin Oncol. 2003 Jul 15;21(14):2636-44. doi: 10.1200/JCO.2003.11.136. PMID 12860938
- [Result] Ceresoli GL, Aerts JG, Dziadziuszko R, Ramlau R, Cedres S, van Meerbeeck JP, Mencoboni M, Planchard D, Chella A, Crino L, Krzakowski M, Russel J, Maconi A, Gianoncelli L, Grosso F. Tumour Treating Fields in combination with pemetrexed and cisplatin or carboplatin as first-line treatment for unresectable malignant pleural mesothelioma (STELLAR): a multicentre, single-arm phase 2 trial. Lancet Oncol. 2019 Dec;20(12):1702-1709. doi: 10.1016/S1470-2045(19)30532-7. Epub 2019 Oct 15. PMID 31628016
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Toms SA, Kim CY, Nicholas G, Ram Z. Increased compliance with tumor treating fields therapy is prognostic for improved survival in the treatment of glioblastoma: a subgroup analysis of the EF-14 phase III trial. J Neurooncol. 2019 Jan;141(2):467-473. doi: 10.1007/s11060-018-03057-z. Epub 2018 Dec 1. PMID 30506499
- [Result] Mrugala MM, Engelhard HH, Dinh Tran D, Kew Y, Cavaliere R, Villano JL, Annenelie Bota D, Rudnick J, Love Sumrall A, Zhu JJ, Butowski N. Clinical practice experience with NovoTTF-100A system for glioblastoma: The Patient Registry Dataset (PRiDe). Semin Oncol. 2014 Oct;41 Suppl 6:S4-S13. doi: 10.1053/j.seminoncol.2014.09.010. Epub 2014 Sep 16. PMID 25213869
- [Result] Kanner AA, Wong ET, Villano JL, Ram Z; EF-11 Investigators. Post Hoc analyses of intention-to-treat population in phase III comparison of NovoTTF-100A system versus best physician's choice chemotherapy. Semin Oncol. 2014 Oct;41 Suppl 6:S25-34. doi: 10.1053/j.seminoncol.2014.09.008. Epub 2014 Sep 16. PMID 25213871
- [Result] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869